CLINICAL TRIAL: NCT02550535
Title: Single Arm Phase I/II Study of the Safety and Efficacy of Gene-modified WT1 TCR Therapy in Patients With Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukaemia (AML) Who Have Failed to Achieve or Maintain an IWG Response Following Hypomethylating Agent Therapy
Brief Title: A Phase I/II Study of Gene-modified WT1 TCR Therapy in MDS & AML Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Medica Ltd (Industry)
Collaborators: University College, London (Other); Cell Therapy Catapult (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-00272-CT2014002
Record Dates: First submitted 2015-04-28; First posted 2015-09-15 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Myelodysplastic Syndromes (MDS); Acute Myeloid Leukaemia (AML)
Keywords: Gene Therapy; WT1 TCR; Gene modified T cels
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gene-modified WT1 TCR-transduced T cells (Experimental): A single dose of bulk WT1 TCR-transduced T cells (≤ 2 x 107/kg) will be intravenously (i.v.) administered following protocol-specified lymphodepletive conditioning regimen. Additionally, daily IL-2 subcutaneous injections (1x106 units/m2 subcutaneously (s.c.)) will be administered for 5 days concomitantly to each subject, following infusion of the ATIMP.
  Interventions: Genetic: Autologous WT1 TCR transduced T cells

INTERVENTIONS:
Genetic: Autologous WT1 TCR transduced T cells — Gene therapy: Autologous WT1 TCR transduced T cells administered by intravenous infusion

SUMMARY:
This is a Phase I/II trial to determine safety, clinical efficacy and feasibility of a gene-modified WT1 TCR therapy in patients with myelodysplastic syndrome (MDS) and acute myeloid leukaemia (AML).

Patient's white blood cells (T cells) will be modified by transferring a gene which enables them to make a new T cell receptor (TCR) that can recognize fragments of a protein called WT1 (Wilms' tumour 1) which is present at abnormally high levels on the surface of myelodysplastic and leukaemic cells.

In this trial, approximately 25 participants with an Human Leukocyte Antigen A2 (HLA-A*0201) tissue type who have failed to achieve or maintain an IWG defined response following hypomethylating agent therapy will be recruited.

DETAILED DESCRIPTION:
This is a Phase I/II trial to determine safety, clinical efficacy and feasibility of a gene-modified WT1 TCR therapy. Following provision of informed consent, each subject will undergo screening assessments, including HLA-A*0201 screening (if not already documented) and a bone marrow aspirate/biopsy (BMA) to determine subject eligibility for the trial.

Subjects will undergo leukapheresis within 14 days of screening.

Once successful manufacture of the WT1 TCR-transduced T cells has been confirmed by the Sponsor, each subject will be administered a lymphodepletive conditioning regimen for five days consisting of fludarabine x 5 days 30mg/m2 intravenous (i.v.) and methylprednisolone x 1 day 500 mg i.v. Upon completion of the conditioning regimen, subjects will receive an infusion of WT1 TCR-transduced T cells of ≤2 x 107/kg, followed by daily IL-2 subcutaneous injections (1 x 106 units/m2 subcutaneous (s.c.) od) for 5 days.

If an IWG response has not been reported (one or more criteria met) at 3 months post-infusion then, if agreed by both the Investigator and Sponsor, the subject will be offered to have a repeat infusion of WT1 TCR-transduced T cells.

Following infusion, subjects will enter an intensive period of out-patient follow-up to observe them for any acute complications and toxicities. Subjects will then be followed monthly in the clinic for the first 6 months for routine safety and clinical evaluations, including disease response evaluations. All subjects will be followed-up for a minimum of 12 months.

ELIGIBILITY:
Key Inclusion criteria:

* The trial will recruit subjects with MDS or AML who have received hypomethylating agent therapy (at least 6 cycles of azacitidine or 4 cycles of decitabine), and are EITHER:
* Relapsed, defined as failing to maintain an initial IWG response

OR

• Stable, defined as failing to achieve an IWG response

Subjects who have received hypomethylating agent therapy as part of a combination regimen may be eligible after discussion with the Sponsor.

1. Subjects aged 18 years or older who have a diagnosis of, EITHER:

   * MDS with an IPSS of intermediate -2, or high and one of the following FAB types:

     * Refractory anaemia with excess blasts (RAEB)
     * Chronic myelomonocytic leukaemia (CMML) with at least 10% bone marrow blasts (WHO CMML II) OR
   * AML (diagnosed according to WHO classification 2008 revision)
2. Subjects with documented HLA-A*0201 positive serotype
3. Subjects with less than 30 per cent bone marrow blasts
4. Subjects with relapsed disease must have less than 5 per cent peripheral blasts
5. Subjects with stable disease must have less than 10 per cent peripheral blasts
6. Subjects with less than a doubling of bone marrow blast count between the start of hypomethylating agent therapy and the date of screening
7. Subjects to complete screen 1 visit within a minimum of 28 days and maximum of 90 days since completion of azacitidine or decitabine therapy. Subjects who have exceeded the 90 day window may be eligible after discussion with the Sponsor.
8. Subjects with ECOG status 0, 1 or 2
9. Subjects who have at least one cytopenia (ANC <1000/μL, platelet count <75,000/μL, Hgb <11g/dL or RBC transfusion dependence)

Key Exclusion criteria:

improvement or molecular response following azacitidine treatment

* CMML patients who have a white blood cell count > 13 x 109/L
* Acute promyelocytic leukaemia (FAB M3 Classification)
* Uncontrolled intercurrent illness
* Active malignancy, except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C virus (HCV) or Hepatitis B virus (HBV) or positive for Human T-Lymphocyte Virus (HTLV) or Syphilis. • Active auto-immune disease
* Clinically significant non-hematologic toxicity after prior therapy chemotherapy higher than grade 1 per Common Terminology Criteria for Adverse Events (CTCAE) (v 4.0)
* Subjects who require haemodialysis or peritoneal dialysis
* Pregnant and lactating women
* Subjects unwilling or unable to use adequate contraceptive precautions at screening and throughout the trial
* Subjects who have undergone major surgery without full recovery within last 28 days prior to screening
* Subjects with known hypersensitivity to cyclophosphamide, fludarabine, methylprednisolone or IL-2 (Interleukin-2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Safety following gene-modified WT1 TCR T cell therapy as measured by suspected unexpected serious adverse reactions (SUSARS) | 12 Months
Proportion of subjects achieving one or more IWG response criteria following gene-modified WT1 TCR T cell therapy | 12 Months

SECONDARY OUTCOMES:
Safety and tolerability of gene-modified WT1 TCR therapy as measured by clinical laboratory parameters and adverse events | 12 Months
Efficacy of WT1 TCR therapy as measured by haematological improvement, overall remission rate, marrow remission, cytogenetic response, molecular response, stable disease, AML transformation, progression free, event free and overall survival | 12 Months
  Haematologic Response (peripheral blood): Haematological response will be assessed by haematology results and capturing data on number of RBC/platelet transfusions given to the subject.
  Marrow Response: Bone marrow aspirate and/or biopsy morphology results will be recorded and assessed for marrow response in combination with peripheral blood response Cytogenetic response: cytogenetic evaluations will be performed on bone marrow aspirates/biopsies obtained during the trial.
  Molecular response: molecular profile evaluations will be performed on bone marrow aspirates/biopsies obtained during the trial.
  Disease response: Investigator will determine response (CR, PR, stable disease (SD), PD/TF) to administration of WT1 transduced T cells based on bone marrow blast count and peripheral blood assessments.
  Subject disease events, progression and survival will be reviewed, assessed and recorded by the Investigator.
Technical feasibility of gene-modified WT1 TCR therapy in subjects with Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukaemia (AML). | 12 Months
Persistence of WT1 TCR-transduced T cells | 12 Months
  Persistence of infused WT1 TCR-transduced T cells by Vβ2.1 and tetramer staining and PCR for Vβ2.1 and TCR-vector fragments.
Functionality and phenotype of WT1 TCR-transduced T cells | 12 Months
  Function will be evaluated by measuring antigen-specific intracellular cytokine production in response to target cells that express HLA-A*201 alleles as well as WT1. Surface differentiation and memory phenotype will be determined using multi-parameter flow cytometry.
WT1 Transcript analysis in AML/MDS cells | 12 Months
  WT1 overexpression will be used as a measure of disease monitoring on peripheral blood and BMA samples. RT-qPCR will be used to detect WT1 transcripts.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Morris, MD, Principal Investigator — University College London Hospitals
Locations (6):
- Belgium (2):
  - AZ St Jan Brugge-Oostende AV, Bruges
  - UZ Leuven, Leuven
- Uniklinikum Dresden, Dresden, Germany
- United Kingdom (3):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - University College London Hospitals NHS Trust, London